CLINICAL TRIAL: NCT00706732
Title: A Single-Site, Phase I/II, Double Blinded, Safety and Immunogenicity Trial of an Alphavirus Replicon Vaccine Expressing Influenza A/Wyoming/03/2003 Hemagglutinin (AVX502) in Adult Volunteers 65 Years of Age or Older
Brief Title: A Safety and Immunogenicity Trial in Adults 65 Years of Age or Over to Prevent Influenza
Acronym: AVX502-003
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AVX502-003
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: Influenza; Flu; A/Wyoming/03/2003; Alphavirus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- T1 (Active Comparator)
  Interventions: Biological: AVX502
- T2 (Active Comparator)
  Interventions: Biological: AVX502
- C1 (Placebo Comparator)
  Interventions: Biological: Placebo
- C2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AVX502 — 2 doses at 2e8 IU given at T=0 and T=4 weeks via the IM route
  Arms: T1
Biological: AVX502 — 2 doses at 2e8 IU given at T=0 and T=4 weeks given via the SC route
  Arms: T2
Biological: Placebo — 2 doses of placebo given at T=0 and T=4 weeks via the IM route
  Arms: C1
Biological: Placebo — 2 doses of placebo given at T=0 and T=4 weeks via the SC route
  Arms: C2

SUMMARY:
The objective of this study is to evaluate the safety of the vaccine and the immune response to the vaccine in healthy adult volunteers 65 years of age or older. Volunteers will be assigned by randomization to receive either the vaccine or an inactive substance (placebo) by injections in the arm on two occasions over one month. The study will last approximately 10 months and will have a total of 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years of age or older
* Good general health without significant physical examination findings or clinically significant abnormal laboratory results
* Available to participate for entire study period
* Acceptable laboratory parameters
* Willingness to have blood stored for up to 10 years for use in additional assays to evaluate immune responses to influenza or the alphavirus vector if such assays become available
* Willingness to refrain from donating blood while participating in the study
* Willingness to delay receipt of 2008-2009 licensed influenza vaccination until after completing study visit 6 procedures (study week 8)
* Signed inform consent obtained before screening and before enrollment

Exclusion Criteria:

* Venous access deemed inadequate for th phlebotomy demands of the study
* Receipt of any other vaccine within 30 days prior to enrollment
* Use of any investigational agent within 30 days prior to enrollment
* Receipt of immunoglobulin or other blood products within 60 days prior to enrollment
* Use of cytotoxic medications within 6 months prior to enrollment
* Use of systemic corticosteroids within 6 months prior to enrollment (except that participants who have completed a course of prednisone, at up to 20 mg per day for up to 7 days, at least 1 month prior to enrollment are eligible for enrollment)
* History of serious adverse reactions to any vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, or abdominal pain
* History of autoimmune disease or splenectomy
* History of malignancy within the last 3 years (except that participants with a diagnosis of basal cell carcinoma of the skin are eligible for enrollment)
* Psychiatric condition that may interfere with the ability to comply with the protocol requirements or to understand informed consent. Specifically excluded are persons with history of psychosis within the past 3 years or history of suicidal attempt or gesture within the past 3 years.
* History of medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* Any condition which leads the investigator to believe that the particpant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for further participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of AVX502 in healthy adult volunteers 65 years of age or older via the frequency of systemic reactogenicity events, local vaccine reactions and Adverse Events | 28 weeks

SECONDARY OUTCOMES:
Evaluate the immunogenicity of AVX502 in healthy adult volunteers 65 years of age and older via serum antibody concentration | 4 weeks after second dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olmsted, Ph.D., Principal Investigator — AlphaVax, Inc.
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

REFERENCES:
- See also: AlphaVax, Inc. — http://www.alphavax.com
- See also: Johnson County Clin-Trials — http://www.jcct.com